CLINICAL TRIAL: NCT05340504
Title: Experimentally Evaluating the Hypothesized Mechanism of Action of N-acetylcysteine for Bipolar Disorder
Brief Title: Evaluating the Hypothesized Mechanism of Action of N-acetylcysteine for Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Milken Institute (Other)
Responsible Party: Principal Investigator, James J. Prisciandaro, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 00117736
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: Bipolar Disorder; Bipolar I Disorder; Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: N-Acetylcysteine, then Washout, then Placebo Oral Capsule (Experimental): Group A will receive NAC 2 times a day for a total of 14 days. On Day 14 they will have a Magnetic Resonance Imaging (MRI) exam. They will then have a 14 day washout period. They will then receive Placebo Oral Capsule 2 times a day for 14 days and have another MRI exam on day 14.
  Interventions: Drug: N-Acetyl cysteine; Drug: Placebo
- Group B: Placebo Oral Capsule, then Washout, then N-Acetylcysteine (Experimental): Group A will receive Placebo Oral Capsule 2 times a day for a total of 14 days. On Day 14 they will have a Magnetic Resonance Imaging (MRI) exam. They will then have a 14 day washout period. They will then receive NAC 2 times a day for 14 days and have another MRI exam on day 14.
  Interventions: Drug: N-Acetyl cysteine; Drug: Placebo

INTERVENTIONS:
Drug: N-Acetyl cysteine — Group A and Group B will receive N-Acetylcysteine (NAC). Group A will receive NAC as their first 14 day condition and Group B will receive NAC as their second 14 day condition. Participants will take NAC for 14 days and then have a MRI exam after completing various assessments (clinical interview, questionnaires, etc).
Drug: Placebo — Group A and Group B will receive Placebo. Group A will receive Placebo as their first 14 day condition and Group B will receive Placebo as their second 14 day condition. Participants will take Placebo Oral Capsule for 14 days and then have a MRI exam after completing various assessments (clinical interview, questionnaires, etc).

SUMMARY:
This research study evaluates the effects of anFDA-approved medication NAC in individuals with Bipolar Disorder. Participants in the study will will be assigned to two medication conditions and will take both NAC and a matched placebo. The order in which they take each medication will be random. Study medication will be taken for 14 days. There will be 5 study visits, with 2 MRI brain imaging scans completed. Questionnaires and clinical interview measures will be completed at study visits along with consistent assessment of potential side effects from study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-60 years
2. Meet DSM-5 criteria for bipolar I or II disorder
3. Able to provide informed consent and read, understand, and accurately complete assessment instruments
4. Willing to commit to medication treatment and follow-up assessments
5. Meets DSM-5 criteria for any mood episode (i.e., Major Depressive, Hypomanic, Manic), Current or In Partial Remission
6. Prescribed daily use of at least one FDA-approved mood stabilizing medication (i.e., lithium, divalproex sodium, lamotrigine, 2nd generation antipsychotic)
7. Willing to abstain from antioxidant supplements (e.g., coenzyme Q-10, vitamin E) for the duration of the study.

Exclusion Criteria:

1. A primary psychiatric diagnosis other than BD (e.g., Schizophrenia)
2. Meet DSM-5 criteria for substance use disorder (other than Tobacco Use Disorder) within the past 6 months.
3. Any uncontrolled neurological condition (e.g., epilepsy) that could confound the results of the study
4. Any history of brain injury with loss of consciousness greater than 5 minutes
5. Any history of mental retardation, dementia, or recent electroconvulsive therapy (in the past 3 months)
6. Any uncontrolled medical condition that may adversely affect the conduct of the study or jeopardize the safety of the participant
7. Hepatocellular disease as indicated by plasma levels of liver transaminases (aspartate transaminase, alanine transaminase) greater than 3 times the normal range
8. Renal insufficiency as indicated by plasma levels of creatinine greater than 2 times the normal range
9. Concomitant use of nitroglycerine, carbamazepine, or any other medication deemed to be hazardous if taken with N-Acetylcysteine (NAC).
10. Medication dose changes of ≥ 20% ≤ 2 weeks prior to testing
11. Women of childbearing potential who are pregnant, lactating, or refuse adequate forms of contraception
12. Current suicidal or homicidal risk
13. Baseline scores greater than 35 on the Montgomery-Asberg Depression Rating Scale or greater than 25 on the Young Mania Rating Scale
14. Has taken NAC in the last month or experienced adverse effects/allergic reaction from it at any time
15. Significant claustrophobia and/or past negative experiences with MRI
16. Presence of non-MRI safe materials in the body (e.g., ferrous metal implants, pacemaker)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Prisciandaro, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University Of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: N-Acetylcysteine, Washout, Then Placebo Oral Capsule: Two, 2-week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), maximum dose of NAC (i.e., 3g/day NAC) (Days 1-14), MRI (Day 14) and medication washout (Day 15-28).
  N-Acetylcysteine: 14 day trial of 3g NAC.
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), maximum dose of matched Placebo Oral Capsule (Days 1-14), and MRI (Day 14).
  Placebo Oral Capsule: 14 day trial of matched placebo.
- Group B: Placebo Oral Capsule, Washout, Then N-Acetylcysteine: Two, 2-week conditions.
  Week 1 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), maximum dose of matched Placebo Oral Capsule (Days 1-14), MRI (Day 14) and medication washout (Day 15-28).
  Placebo Oral Capsule: 14 day trial of matched placebo.
  Week 2 condition will consist of an in-person study visit for assessment and dispensing of medication (Day 1), maximum dose of NAC (i.e., 3g/day NAC) (Days 1-14), and MRI (Day 14).
  N-Acetylcysteine: 14 day trial of 3g NAC.
Period: Overall Study
Arm/Group | Group A: N-Acetylcysteine, Washout, Then Placebo Oral Capsule | Group B: Placebo Oral Capsule, Washout, Then N-Acetylcysteine
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: N-Acetylcysteine, Washout, Then Placebo Oral Capsule | Group B: Placebo Oral Capsule, Washout, Then N-Acetylcysteine | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34.5 [20 to 55] | 41.33 [24 to 60] | 37.92 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 5 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in dACC GSH Levels Through Proton Magnetic Resonance Spectroscopy
Description: Brain GSH levels, balanced with water and CSF-corrected, in dorsal anterior cingulate measured via Proton Magnetic Resonance Spectroscopy
Time Frame: Day 14 of each experimental condition
Population: Overall number of participants analyzed includes participants who completed full study protocol (i.e. 2, 2-week medication trials and 1, 2-week washout period). Two participants have been removed from outcome measure data (1 - participant lost to follow up and did not complete placebo condition, 1 - participant's MRI data was unusable due to excessive head motion). Data from these 2 participants has been included in other portions of this study record (Adverse Events, Demographics, etc).
Measure: Mean (Standard Deviation); unit: Institutional Units
Groups:
- N-Acetylcysteine: N-Acetylcysteine: 14 day trial of N-Acetylcysteine (3g/day) followed by MRI (Day 14)
- Placebo: Placebo: 14 day trial of matched Placebo Oral Capsule followed by MRI (Day 14)
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 10 | 10
Institutional Units | 2.426 (0.341) | 2.207 (0.423)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected over each participant's total study duration. This duration was a 6-week period for each participant (i.e., 2, 2-week condition periods separated by 1, 2-week washout period). Adverse event data collection took place for the entirety of the study which was 1 year.
Description: At each study visit following the initial screening visit, study participants were assessed by the study medical doctor for any adverse events. Adverse events were recorded, rated on a severity scale, determined their relation to the study medication, and any treatment or intervention needed was discussed. The study medical doctor followed up with all previously reported adverse events at the following visits to determine if the events had ceased.
Groups:
- N-Acetylcysteine: N-Acetylcysteine: 14 day trial of N-acetylcysteine 3g/day
- Placebo Oral Tablet: Placebo Oral Tablet: 14 day trial of matched placebo
- Washout: Washout: 14 day washout period from study medications
Arm/Group | N-Acetylcysteine | Placebo Oral Tablet | Washout
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/11 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=12) | Placebo Oral Tablet (N=11) | Washout (N=12)
Skin Growth (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT05340504/Prot_SAP_000.pdf